CLINICAL TRIAL: NCT03856320
Title: A Randomized Pilot Study of a Video-based Obesity Educational Intervention (CDA 15-060)
Brief Title: Teaching Obesity Treatment Options to Adult Learners Trial
Acronym: TOTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The Clowes Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDX 18-001
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Patient Education; Weight Loss
Keywords: Obesity; Patient Education; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: An educational video describing obesity treatment options available in the VA.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the patient's allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patient attends a MOVE! visit (weight management visit).
- Intervention (Experimental): Patient attends a MOVE! visit (weight management visit) and watches an educational video describing obesity treatment options available in the VA.
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: Educational Video — An educational video describing obesity treatment options available in the VA.
  Arms: Intervention

SUMMARY:
Obesity is the second leading cause of death in the U.S. The treatment of obesity and its related health issues, including cardiovascular disease and diabetes, exceeds $150 billion annually. "Morbidly" or "severely" obese patients - defined by a body mass index [BMI] of >35 kg/m2 or greater - are especially high risk for serious complications due to their weight. Within the Veterans Health Administration (VA) system, nearly 600,000 patients are severely obese. These Veterans create significant costs for the VA system, experience poorer quality of life, and have shortened lifespans. Bariatric surgery is the most effective treatment for severe obesity for weight loss, resolving weight-related health issues, and quality of life. Bariatric surgery is supported as a treatment option by many national societies, including those representing primary care and endocrinology. However, less than 1% of Veterans who qualify for bariatric surgery undergo it. Reasons for low utilization are unclear, although the investigators' preliminary research suggests that there are various patient, provider and system level barriers to severe obesity care. The goal of this study is to pilot-test an educational video that aligns patient preferences with treatment options to improve the care that severely obese Veterans receive.

DETAILED DESCRIPTION:
Obesity is the second leading cause of death in the U.S. The treatment of obesity and its related comorbidities, including cardiovascular disease and diabetes, exceeds $150 billion annually. "Morbidly" or "severely" obese patients - defined by a body mass index [BMI] of >35 kg/m2 or greater - are especially high risk for serious complications due to the metabolic and physiologic derangements that occur with severe obesity. Within the Veterans Health Administration (VA) system, nearly 600,000 patients are severely obese. These Veterans exert significant costs on the VA system, experience poorer quality of life, and have shortened lifespans. Bariatric surgery is the most effective treatment for severe obesity for weight loss, comorbidity resolution, and quality of life. Bariatric surgery is supported as a treatment option by many national societies, including those representing primary care and endocrinology. However, less than 1% of Veterans who qualify for bariatric surgery undergo it. Reasons for low utilization are unclear, although the investigators' preliminary research suggests that there are various patient, provider and system level barriers to severe obesity care. The goal of this study is to pilot-test an educational video that aligns patient preferences with treatment options to optimize the care that severely obese Veterans receive.

ELIGIBILITY:
Inclusion Criteria:

* Veterans scheduled to attend an in-person MOVE! visit led by a dietitian at the main VA hospital.

Exclusion Criteria:

* No access to telephone, doesn't speak English as their primary language, has undergone bariatric surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke M Funk, MD MPH, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Funk LM, Breuer CR, Venkatesh M, Muraveva A, Alagoz E, Hanlon BM, Raffa SD, Voils CI. Protocol and short-term results for a feasibility randomized controlled trial of a video intervention for Veterans with obesity: The TOTAL (Teaching Obesity Treatment Options to Adult Learners) pilot study. Contemp Clin Trials Commun. 2021 Jun 29;23:100816. doi: 10.1016/j.conctc.2021.100816. eCollection 2021 Sep. PMID 34258469

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 20 | 22
Completed | 20 | 20
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.1) | 60.7 (10.9) | 59.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 18 | 19 | 37
  Black, non-Hispanic | 0 | 0 | 0
  Hispanic | 0 | 1 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
BMI [Mean (Standard Deviation); unit: kg/m^2] | 40.7 (7.8) | 43.1 (5.3) | 41.9 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: The proportion of patients who were contacted by the study team who also consented and provided baseline assessment data.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- All Attempted Recruitment: # of participants randomized to the study divided by # of participants sent a recruitment letter
Arm/Group | All Attempted Recruitment
Number analyzed (Participants) | 89
Participants | 42

2. Primary Outcome: Retention
Description: The proportion of patients who consented and completed the baseline assessment who also completed the post assessment.
Time Frame: 7-14 days
Measure: Count of Participants; unit: Participants
Groups:
- Retention: # of participants who completed the one-week post-intervention assessment divided by # of participants who were randomized.
Arm/Group | Retention
Number analyzed (Participants) | 42
Participants | 40

ADVERSE EVENTS:
Time Frame: Approximately 9 months
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03856320/Prot_SAP_000.pdf